CLINICAL TRIAL: NCT04316481
Title: ALERTS Continued Access Study- IDE G060259 Supplement
Brief Title: IDE-ALERTS Continued Access Study
Acronym: ALERTS-CAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA Approval was received for the Model AMSG3-E IMD and therefore commercial implants could be started. There was no longer any need to implant under the CAS. CAS patients were transitioned to commercial patients.
Sponsor: Angel Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WRB 1281733
Record Dates: First submitted 2020-03-12; First posted 2020-03-20 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: Continued Access
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AngelMed Guardian System (Other): All eligible subjects will have the AngelMed Guardian System implanted with alerting features turned ON; receive an external device which provides additional alerting; and receive training on system use.
  Interventions: Device: AngelMed Guardian System

INTERVENTIONS:
Device: AngelMed Guardian System — The AngelMed Guardian System detects potential ongoing ACS events, characterized by sustained ST segment changes, and alerts the patient to seek medical attention for those potential ACS events. The Guardian System is indicated as an adjunct to patient recognized symptoms.

SUMMARY:
This Continued Access IDE Study includes a subset of former ALERTS trial (NCT00781118) patients and provides performance data for a refined Guardian implantable medical device (AMSG3-E) with a new battery designed to extend device longevity.

DETAILED DESCRIPTION:
This Continued Access IDE Study is a prospective, non-randomized, multi-center (up to 25 sites) study designed to provide performance assessment of a refined Guardian implantable medical device (AMSG3-E) through controlled access of a replacement Guardian System to a subset of former ALERTS patients while waiting for FDA approval of the AMSG3-E. The AMSG3-E contains a drop-in replacement battery designed to extend the life of the implant to potentially exceed the previous 3-years implant life. Eligible patients will include those that exited the ALERTS study and chose to leave the device and/or lead in place. Eligible patients must also continue to meet ALERTS inclusion criteria and not have developed any exclusion criteria since exiting the ALERTS study.

ELIGIBILITY:
Inclusion Criteria (all must be true):

* Subject previously participated in the ALERTS study and currently has either a Guardian System IMD plus IS-1 lead or IS-1 lead still in place and hasn't developed exclusion criteria.
* Subject (men or women) is at least 21 years of age.
* Women of childbearing age must have a negative pregnancy test or confirmation of one of the following:

  1. Post-menopause or amenorrhoeic during the past year
  2. Surgical sterilization
  3. Use of effective contraceptive method

Exclusion Criteria:

* In the investigator's opinion, subject lacks ability to respond appropriately to alarms, e.g., illiteracy, poor memory or cognitive function, dementia or other condition affecting memory function, etc.
* Known compromised tissue at the site of lead implantation in the apex of the right ventricle, e.g., prior infarct affecting the RV apex location.
* A permanent pacemaker or ICD is already in place or the patient is indicated for ICD or pacemaker implantation based on the guidelines published by the American College of Cardiology as Class I and IIa recommendations. Class IIb recommendations are at the investigator's discretion.
* Subject cannot feel the IMD vibration when placed on top of the skin on the left pectoral side of the chest.
* Subject has recurrent or persistent atrial fibrillation.
* Subject has recurrent or persistent non-sinus cardiac rhythm, second- or third-degree atrioventricular blocks, QRS duration greater than 120 ms, Benign Early Repolarization (BER), Brugada Syndrome, (LBB, BBB, RBB) or Rate Induced BBB.
* Subject has left ventricular hypertrophy evidenced by EKG criteria.
* Subject has any condition preventing the subcutaneous implantation of the Guardian System in a left pectoral pouch, such as:

  1. superior vena cava thrombosis,
  2. subcutaneous tissue deemed inappropriate for the procedure
  3. prior central venous access via portacath, Hickman, Groshong, or similar placed in a left pectoral location or left side PICC line.
* Extremely heavy alcohol consumption (participates in binge drinking that leads to alcohol intoxication) or has history of alcohol or illicit drug abuse within past 5 years.
* Evidence of unresolved infection (fever > 38o C and/or leukocytosis > 15,000).
* History of bleeding disorders or severe coagulopathy (platelets < 100,000 plts/ml; APTT or PT > 1.3 x reference range).
* Subject has had a hemorrhagic stroke or transient ischemic attack (TIA) in the past 6 months.
* Subject has other severe diseases, such as cancer or refractory congestive heart failure, associated with limitation of life expectancy (less than 1 year), which may lead to inadequate compliance to the protocol or confusing data interpretation.
* Subject has clinical conditions such as heart diseases, difficult-to-control blood pressure, difficult-to-control insulin-dependent diabetes or serious prior infections attributed to the diabetes, or others that, at the investigator's discretion, could seriously affect the subject's current clinical condition during study procedures.
* Subject has current participation or previous participation in another drug or device study in the past 30 days that conflicts with this study as determined by the study sponsor.
* Gastro-intestinal hemorrhage in the past 6 months.
* Subject has any situation in which the use of aspirin is contraindicated for at least 6 months.
* Subject has epilepsy
* Subject has known severe allergies, e.g., peanut, bee sting.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Rate of Serious Adverse Events (SAE) | 5 years
  Annual rate of SAEs related to the device or procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell W Krucoff, MD, Principal Investigator — Duke University
Locations (1):
- Orange County Heart Institute and Research Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gibson CM, Holmes D, Mikdadi G, Presser D, Wohns D, Yee MK, Kaplan A, Ciuffo A, Eberly AL 3rd, Iteld B, Krucoff MW. Implantable Cardiac Alert System for Early Recognition of ST-Segment Elevation Myocardial Infarction. J Am Coll Cardiol. 2019 Apr 23;73(15):1919-1927. doi: 10.1016/j.jacc.2019.01.014. Epub 2019 Mar 3. PMID 30842028
- [Result] Holmes DR Jr, Krucoff MW, Mullin C, Mikdadi G, Presser D, Wohns D, Kaplan A, Ciuffo A, Eberly AL 3rd, Iteld B, Fischell DR, Fischell T, Keenan D, John MS, Gibson CM. Implanted Monitor Alerting to Reduce Treatment Delay in Patients With Acute Coronary Syndrome Events. J Am Coll Cardiol. 2019 Oct 22;74(16):2047-2055. doi: 10.1016/j.jacc.2019.07.084. PMID 31623762
- [Result] Kazmi SHA, Datta S, Chi G, Nafee T, Yee M, Kalia A, Sharfaei S, Shojaei F, Mirwais S, Gibson CM. The AngelMed Guardian(R) System in the Detection of Coronary Artery Occlusion: Current Perspectives. Med Devices (Auckl). 2020 Jan 7;13:1-12. doi: 10.2147/MDER.S219865. eCollection 2020. PMID 32021496
- See also: SSED — https://www.accessdata.fda.gov/cdrh_docs/pdf15/P150009B.pdf